CLINICAL TRIAL: NCT00872937
Title: Retrospective Study of the Relationship Between Human Papillomavirus Genotype and Cervical Epithelial Lesions
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 200812138R
Record Dates: First submitted 2009-03-30; First posted 2009-03-31 (Estimated); Last update posted 2012-05-17 (Estimated); Status verified 2012-03

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Human papillomavirus (HPV) infection plays a key role in the carcinogenesis of cervical cancer and pre-invasive lesions. There are hundred types of HPV, including high risk and low risk types, and it is proved the close association between the cervical cancer and high risk HPV. While HPV 16 and 18 are known to be the leading two genotypes detected in women with cervical neoplasm worldwide, there is considerable difference in the other prevalent high risk genotypes in different geographic areas. It is important to establish the local database about the cervical intraepithelial lesions and the related prevalent HPV genotypes. The investigators designed a retrospective study which included total 784 patients managed at our hospital from January 1, 2000 to December 31, 2007. The present study was to investigate the HPV genotypes in the Taiwanese female patients with abnormal cervical cytology and analyses the association between HPV types and cervical pre-invasive lesions. It could provide the guide for the clinicians in the management of patients with abnormal cytological change of Pap smear.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* People infected with HPV type 16 but without CIN lesions
* Patients with CIN lesions
* Patients with cervical cancer from National Taiwan University Hospital
* Informed consent is obtained, and the protocols are reviewed and approved by the appropriate Investigative Review Boards.

Exclusion Criteria:

* None

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: cervical cancer patients with HPVinfection
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2009-03; Primary Completion 2009-03 (Actual); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
overall survival | from disease diagnosis to death

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Fang Cheng, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan